CLINICAL TRIAL: NCT06340867
Title: Effect of Two Different Intraoral Scanners on the Scanning Quality and Time in Patients With/Without Orthodontic Brackets
Brief Title: Intraoral Scanner With and Without Orthodontic Brackets
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdulrahman Majed Ahmed Joureyah, master degree student, Faculty of Dentistry , Cairo university, Cairo University
Other Study IDs: 30723
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Intra-oral Scanner; Adolescent Behavior
Keywords: Dentsply with/ without bracket
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CEREC primescan intra-oral scanner — intra-oral scanner

SUMMARY:
this study aim to evaluate the effect of two different intraoral scanners on the scanning Quality and Time in Patients With/Without Orthodontic Brackets

DETAILED DESCRIPTION:
aim of study : evaluate two types of Intra-oral scanner in patients with/without orthodontics brackets

methodology:

* patient preparation diagnosis, photos, x-rays
* starting scanning in 3 techniques bucco-palatal , palato-buccal ,s shape
* brackets bonding by indirect technique
* scanning after brackets placement also by same 3 techniques
* data measurements by linear and angular measurements.

outcome:2 scanners will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes.
2. Full permanent dentition cases.
3. Class I/II/III molar relationship.
4. Mild to moderate crowding cases

Exclusion Criteria:

1. Dental anomalies.
2. Congenital missing teeth.
3. Impaction.
4. Orthognathic surgery

Ages: 14 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: full permenant dentition with mild to moderate crowding
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
compare the readings resulted from the models produced from the 3 scanners (2 intraoral scanners + the desktop scanner) before bonding and to compare the 2 intraoral scanners after bonding. | 3 to 4 weeks
  using 3 techniques Bucco-palatal, Palato-buccal, S-shape technique collect data and using linear , teeth dimension measurements and angular measurements in 3 shape orthodontic software for data analysis linear measurements will be maxillary/ mandibular inter canine width, maxillary/mandibular inter premolar width , maxillary/mandibular inter molar width , maxillary/ mandibular anterior arch length , maxillary/ mandibular total arch length secondly teeth dimensions by 3shape orthodontic software by measure each tooth from mesial to distal

SECONDARY OUTCOMES:
compare the readings resulted from the models produced from the 2 scanners with and without orthodontic brackets. | 3 to 4 weeks
  measure according to repeatedly scans done by 2 different intra-oral scanners (primescan and carestream) on dental arch using 3 techniques bucco-palatal, palato-buccal and s shape before bonding brackets and after bonding then used 3 shape orthodontic software to superimpose the repeatedly scans on the dental arch either primescan or carestream using ( accuracy and precision) to see if the scans appears clear or deviated with / without brackets

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided